CLINICAL TRIAL: NCT02351791
Title: An Exploratory Study Investigating Human Skin Reaction to Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CP254
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Ileostomy
MeSH Terms: interventions — Sugp2 protein, mouse

ARMS (2):
- Patch 1, 3 and 5 (Experimental): Patch 1, Patch 3 and Patch 5 applied on peristomal skin. Patch 1 - Patch 6 applied on healthy abdominal skin
  Measurements of skin at three locations of each patch: Center and under adhesive.
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: Patch 5; Other: Patch 6
- Patch 2, 4 and 6 (Experimental): Patch 2, Patch 4 and Patch 6 applied on peristomal skin. Patch 1- Patch 6 applied on healthy abdominal skin Measurements of skin at three locations of each patch: Center and under adhesive.
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: Patch 5; Other: Patch 6

INTERVENTIONS:
Other: Patch 1 — Patch 1:standard adhesive with own feces in sleeve
Other: Patch 2 — Patch 2:standard adhesive with own feces mixture in sleeve
Other: Patch 3 — Patch 3: standard adhesive with simulated feces in sleeve
Other: Patch 4 — Patch 4:standard adhesive with simulated feces mixture in sleeve
Other: Patch 5 — Patch 5:standard adhesive with buffer in sleeve
Other: Patch 6 — Patch 6:standard adhesive with buffer mixture in sleeve

SUMMARY:
The primary purpose of the study is to investigate the impact that feces mixtures have on the peristomal skin when using a standard adhesive.

DETAILED DESCRIPTION:
Six types of patches are tested:

Patch 1: Standard adhesive with own feces

Patch 2: Standard adhesive with own feces mixture

Patch 3: Standard adhesive with simulated feces

Patch 4: Standard adhesive with simulated feces mixture

Patch 5: Standard adhesive with buffer (control)

Patch 6: Standard adhesive with buffer feces mixture (control)

Each subject is randomized to one of two arms testing three patches on the peristomal skin (patch 1, 3 and 5 or patch 2, 4 and 6). Furthermore, within each arm an attempt will be made to randomize each of the three patches on the peristomal skin to one of three locations surrounding the stoma (upper left, upper right, lower). On the healthy contralateral abdominal skin the subjects test all six patches.

A run in period with 2 subjects (healthy volunteers) was conducted to clarify the length of the test period. They were exposed to 4 patches (patch 3-6) on healthy abdominal skin which was removed at 2 different time slots. Based on the results the test period was established

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have had an ileostomy for more than one year
* Have normal to slightly red skin on the area used in the evaluation
* Has an ileostomy with a diameter up to (≤) 35 mm
* Have a peristomal area accessible for applied patches (assessed by investigator)

Exclusion Criteria:

* Currently receiving or have within the past 2 months received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment
* Are pregnant or breastfeeding
* Having dermatological problems in the peristomal- or abdominal area (assessed by investigator)
* Participating in other interventional clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, PhD, Principal Investigator — Coloplast A/S
Locations (1):
- Videncenter for Saarheling, Copenhagen NV, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Peristomal Patches: Patch 1, 3 and 5: Patch 1, Patch 3 and Patch 5 applied on peristomal skin. Patch 1 - Patch 6 applied on healthy abdominal skin
  Measurements of skin at three locations of each patch: Center and under adhesive.
  Patch 1: Patch 1:standard adhesive with own feces in sleeve
  Patch 2: Patch 2:standard adhesive with own feces mixture in sleeve
  Patch 3: Patch 3: standard adhesive with simulated feces in sleeve
  Patch 4: Patch 4:standard adhesive with simulated feces mixture in sleeve
  Patch 5: Patch 5:standard adhesive with buffer in sleeve
  Patch 6: Patch 6:standard adhesive with buffer mixture in sleeve
- Peristomal Patches: Patch 2, 4 and 6: Patch 2, Patch 4 and Patch 6 applied on peristomal skin. Patch 1- Patch 6 applied on healthy abdominal skin Measurements of skin at three locations of each patch: Center and under adhesive.
  Patch 1: Patch 1:standard adhesive with own feces in sleeve
  Patch 2: Patch 2:standard adhesive with own feces mixture in sleeve
  Patch 3: Patch 3: standard adhesive with simulated feces in sleeve
  Patch 4: Patch 4:standard adhesive with simulated feces mixture in sleeve
  Patch 5: Patch 5:standard adhesive with buffer in sleeve
  Patch 6: Patch 6:standard adhesive with buffer mixture in sleeve
Period: Overall Study
Arm/Group | Peristomal Patches: Patch 1, 3 and 5 | Peristomal Patches: Patch 2, 4 and 6
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peristomal Patches: Patch 1, 3 and 5 | Peristomal Patches: Patch 2, 4 and 6 | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (12.9) | 64.1 (5.2) | 63.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Trans Epidermal Water Loss After Test of Patches.
Description: Trans Epidermal Water Loss is a standardized non-invasive method for describing the barrier function of the skin. Damage to the skin surface (stratum corneum) will lower the barrier of the skin and thereby increase water loss. This can be used as a measure for the damaging effect of the adhesives to the skin. Trans Epidermal Water Loss is measured by applying a probe to the skin surface and is assessed nine times for each patch after applying the patch: three repeated measurements of the skin covered by the center of the patch (Center), as well as three repeated measurements of the skin covered by the adhesive (Under adhesive).
Time Frame: Approximately 7-10 hours
Population: three repeated measurements per participant were performed and used in analysis e.g. 12 participants have 3x12=36 units analysed.
Measure: Mean (Standard Deviation); unit: g/m^2/h
Units Other Than Participants: 3 repeated measurements per participant
Groups:
- Peristomal Skin Patch 1 Center; Abdominal Skin Patch 1 Center: Measurement on skin (in the center of the patch) exposed to patch 1 (standard adhesive with own feces in sleeve)
- Peristomal Skin Patch 2 Center; Abdominal Skin Patch 2 Center: Measurement on skin (in the center of the patch) exposed to patch 2 (standard adhesive with own feces mixture in sleeve)
- Peristomal Skin Patch 3 Center; Abdominal Skin Patch 3 Center: Measurement on skin (in the center of the patch) exposed to patch 3 (standard adhesive with simulated feces in sleeve)
- Peristomal Skin Patch 4 Center: Measurement on skin (in the center of the patch) exposed to patch 4 (standard adhesive with simualted feces mixture in sleeve)
- Peristomal Skin Patch 5 Center; Abdominal Skin Patch 5 Center: Measurement on skin (in the center of the patch) exposed to patch 5 (standard adhesive with buffer in sleeve)
- Peristomal Skin Patch 6 Center; Abdominal Skin Patch 6 Center: Measurement on skin (in the center of the patch) exposed to patch 6 (standard adhesive with buffer mixture in sleeve)
- Abdominal Skin Patch 4 Center: Measurement on skin (in the center of the patch) exposed to patch 4 (standard adhesive with simulated feces mixture in sleeve)
- Peristomal Skin Patch 1 Under Adhesive; Abdominal Skin Patch 1 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 1 (standard adhesive with own feces in sleeve)
- Peristomal Skin Patch 2 Under Adhesive; Abdominal Skin Patch 2 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 2 (standard adhesive with own feces mixture in sleeve)
- Peristomal Skin Patch 3 Under Adhesive; Abdominal Skin Patch 3 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 3 (standard adhesive with simulated feces in sleeve)
- Peristomal Skin Patch 4 Under Patch: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 4(standard adhesive with simulated feces mixture in sleeve)
- Peristomal Skin Patch 5 Under Adhesive; Abdominal Skin Patch 5 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 5 (standard adhesive with buffer in sleeve)
- Peristomal Skin Patch 6 Under Patch: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 6 (standard adhesive with buffer mixture in sleeve)
- Abdominal Skin Patch 4 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 4 (standard adhesive with simulated feces mixture in sleeve)
- Abdominal Skin Patch 6 Under Adhesive: Measurement on skin (covered by adhesive after removal of patch) exposed to patch 6 (standard adhesive withbuffer mixture in sleeve)
Arm/Group | Peristomal Skin Patch 1 Center | Peristomal Skin Patch 2 Center | Peristomal Skin Patch 3 Center | Peristomal Skin Patch 4 Center | Peristomal Skin Patch 5 Center | Peristomal Skin Patch 6 Center | Abdominal Skin Patch 1 Center | Abdominal Skin Patch 2 Center | Abdominal Skin Patch 3 Center | Abdominal Skin Patch 4 Center | Abdominal Skin Patch 5 Center | Abdominal Skin Patch 6 Center | Peristomal Skin Patch 1 Under Adhesive | Peristomal Skin Patch 2 Under Adhesive | Peristomal Skin Patch 3 Under Adhesive | Peristomal Skin Patch 4 Under Patch | Peristomal Skin Patch 5 Under Adhesive | Peristomal Skin Patch 6 Under Patch | Abdominal Skin Patch 1 Under Adhesive | Abdominal Skin Patch 2 Under Adhesive | Abdominal Skin Patch 3 Under Adhesive | Abdominal Skin Patch 4 Under Adhesive | Abdominal Skin Patch 5 Under Adhesive | Abdominal Skin Patch 6 Under Adhesive
Number analyzed (Participants) | 12 | 10 | 12 | 10 | 12 | 10 | 22 | 22 | 22 | 22 | 22 | 22 | 12 | 10 | 12 | 10 | 12 | 10 | 22 | 22 | 22 | 22 | 22 | 22
Number analyzed (3 repeated measurements per participant) | 36 | 30 | 36 | 30 | 36 | 30 | 66 | 66 | 66 | 66 | 66 | 66 | 36 | 30 | 36 | 30 | 36 | 30 | 66 | 66 | 66 | 66 | 66 | 66
g/m^2/h | 45.8 (29.3) | 22.9 (16.4) | 36.8 (21.7) | 19.6 (11.6) | 15.7 (6.9) | 13.3 (7.1) | 30.1 (25.5) | 22.7 (23.1) | 31.5 (27.7) | 14.5 (12.7) | 13.2 (8.7) | 12.2 (7.6) | 19.5 (16.4) | 12.3 (8.7) | 14.5 (11.7) | 14.7 (7.6) | 13.8 (8.8) | 15.1 (8.1) | 19.0 (12.7) | 19.9 (16.5) | 18.7 (15.4) | 17.3 (15.1) | 15.3 (11.1) | 15.7 (10.4)

ADVERSE EVENTS:
Time Frame: 17 days
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Groups:
- All Participants: This population also includes the two subject who were included in the screening period. Both AEs were related to the investigational procedures (one to the biopsy and one to the pre-stripping of the skin). Thus the AEs are not reported for each intervention separately as the AEs were unrelated to intervention.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=24)
infection in biopsies (Infections and infestations) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — eczema on the pre-stripped abdominal area

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes